CLINICAL TRIAL: NCT02631668
Title: The Efficacy and Safety of Vitamin C for Iron Supplementation Therapy in Adult Patients With Iron Deficiency Anemia(IDA)
Brief Title: the Efficacy and Safety of Vitamin C for Iron Supplementation in Adult IDA Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, xiao-qin wang, professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2015-270
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Anemia, Iron-Deficiency
Keywords: iron deficiency anemia, vitamin C, ferrous succinate
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous succinate; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ferrous succinate and vitamin C (Experimental): In this group, the patients received 100mg ferrous succinate and 200mg vitamin C three times per day for 3-4 months
  Interventions: Drug: ferrous succinate and vitamin C
- ferrous succinate with normal dosage (Active Comparator): In this group, the patients received 100mg ferrous succinate three times per day for 3-4 months
  Interventions: Drug: ferrous succinate
- ferrous succinate with double dosage (Active Comparator): In this group, the patients received 200mg ferrous succinate three times per day for 3-4 months
  Interventions: Drug: ferrous succinate

INTERVENTIONS:
Drug: ferrous succinate and vitamin C — As experimental group, when patients take the tablets of ferrous succinate, they also take vitamin C at the same time
  Arms: ferrous succinate and vitamin C
Drug: ferrous succinate — As active comparator, patients take the tablets of ferrous succinate with normal dosage in clinical practice
  Arms: ferrous succinate with normal dosage
Drug: ferrous succinate — As another active comparator, patients take the tablets of ferrous succinate with double dosage
  Arms: ferrous succinate with double dosage

SUMMARY:
IDA patients ofen receive ferrous succinate treatment to speed up the recovery of anemia, the doctor will prescribe ferrous succinate with or without vitamin C according to their own preferences. In theory, only the divalent iron can be absorbed in duodenum and upper jejunum, vitamin C can oxidize ferric iron into divalent iron and maintains a certain degree of acidity in the intestine, and then promotes the absorption of iron. In current clinical practice, it's lack of randomized controlled trial(RCT) about the efficacy and safety of vitamin C for iron supplementation in patients with IDA. In this study, the efficacy and safety of vitamin C for iron supplementation in adult IDA patients are explored by RCT. The dosage regimens of ferrous succinate with or without vitamin C are randomly assigned to patients who meet the inclusion criteria, and these patients are followed up every two weeks. On the one hand, whether the addition of vitamin C can accelerate the recovery of anemia is evaluated, on the other hand, whether the addition of vitamin C can increase the incidence of gastrointestinal tract discomfort is aslo appraised , the discomfort include vomiting, nausea, abdominal pain, diarrhea and constipation. We hypothesis that vitamin C can increase the absorption of iron and accelerate the recovery of anemia, it also increases incidence of gastrointestinal adverse events because of increased iron absorption at the same time.

DETAILED DESCRIPTION:
BACKGROUND Iron deficiency(ID) causes approximately half of all anemia cases worldwide, a moderate degree of iron-deficiency anemia(IDA) affected approximately 610 million people worldwide or 8.8% of the population. It is slightly more common in female (9.9%) than males (7.8%). In 2013, anemia due to iron deficiency resulted in about 183,000 deaths. IDA is an urgent problem to be solved.

Iron deficiency anemia(IDA) is anemia due to not enough iron. Anemia is defined as a decrease in the amount of red blood cells (RBCs) or hemoglobin in the blood. It is caused by insufficient dietary intake and absorption of iron, or iron loss from bleeding. In babies and adolescents, rapid growth may outpace dietary intake of iron, and result in deficiency without disease or grossly abnormal diet. In women of childbearing age, heavy or long menstrual periods can also cause mild iron-deficiency anemia. Anemia is sometimes treatable, but certain types of anemia may be lifelong. If the cause is dietary iron deficiency, eating more iron-rich foods, such as beans, lentils or red meat, or taking iron supplements will usually correct the anemia.

In clinic, IDA clinically divided into three stages: ID, iron deficiency erythropoiesis (iron deficiency erythropoiesis, IDE) and IDA. The first stage is the reduction of iron storage, and there is a history of inadequate iron absorption; the second stage is the IDE, in addition to iron reduction or lack of external storage, transferrin is also reduced, the intake of iron in red blood cells is reduced compared to normal condition at this time; IDA is the last stage of iron deficiency. If the patients are diagnosed with ID and this condition can be corrected by diet therapy; if it reaches the IDA criteria, it's need to take iron orally and improve symptoms as soon as possible, but the most important is to find the cause of iron deficiency. Ferrous succinate is commonly used to treat IDA in clinic, mainly absorbed in the duodenum and proximal jejunum in the form of ferrous iron. In health people, 5% to 10% of the iron are absorbed after taken orally. the absorption proportion is increased to 20%~30% in IDA patients. After absorbed, ferrous iron can bind to transferrin and enter the blood circulation, and then involve in the production of red blood cells as raw materials. In clinical practice, the doctor will prescribe ferrous succinate with or without vitamin C according to their own preferences. Vitamin C Involves in many biological processes in vivo, such as, collagen formation, tissue repair, the synthesis of phenylalanine, tyrosine, metabolism of folic acid, iron and maintains vascular integrity. Researchers have shown that increased iron intake with vitamin C can prevent anemia,the application of vitamin C can reduce the toxicity symptoms in genotoxic caused by ferric iron, it demonstrates that vitamin C is safe when combined with ferrous succinate. In theory, only the divalent iron can be absorbed in the duodenum and upper jejunum, vitamin C can oxidize ferric iron into divalent iron and maintains a certain degree of acidity in the intestine, and then promotes the absorption of iron. However, the feasibility in theory can not represent the clinical practice. So it's necessary to explore the efficacy and safety of vitamin C for iron supplementation in adult IDA patients through randomized controlled trial(RCT).

PROCEDURE Before the start of this study, the manila envelope is used to carry out the random allocation scheme, different treatment options are randomly loaded into the envelope according to the randomization generated by Stata 11.0 software. In terms of the inclusion criteria, We write the serial number of patients on the envelope after signing informed consent form and give different treatments according to the internal treatment option in envelope. In addition to the above treatment, increased intake of protein, calcium, iron, vitamins and essential fatty acids, appropriate heat are also advised at the same time. In order to check the compliance of the subject, the drug package and aluminum cardboard are asked to return to researchers at follow-up every two weeks, patients should be emphasized that they return all the drug packages, including the pharmaceutical packages that are not taken and run out of, which will help researchers to analyze the patient medication correctly. The number of tablets is to count and determine how much of the remaining drugs and the drugs the patients have taken. During the period of study, patients who participate in this study are not allowed to use other drugs that may affect the effect of iron supplementation. In special circumstances, the patient will be excluded because of using other drugs that affect the absorption of iron or vitamin C. The patients will receive blood routine examination at follow-up every two weeks, the results of examination,the reason and number of termination and loss, the incidence of adverse events in patients, such as, nausea, vomiting, abdominal pain, diarrhea and constipation are all recorded. Finally, we analyze the data to determine the effect and safety of vitamin C for iron supplementation. In this study, we hypothesis that vitamin C can increase the absorption of iron and accelerates the recovery of anemia, it also increases the incidence of gastrointestinal adverse events because of increased iron absorption at the same time.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin (Hb) < 120 g/L in men and Hb < 110 g/L in women; Mean Corpuscular Volume(MCV) < 80 fl, Mean Corpuscular Hemoglobin(MCH) < 27 pg, and Mean Corpuscular Hemoglobin Concentration(MCHC) < 0.32; the blood biochemical examination: serum ferritin < 12 g/L, serum iron < 8.95 mol/L, transferrin saturation <15%, and total iron binding capacity>64.44 mol/L; with a history of Menorrhagia, monophagia or eating disorders; Willing to sign a Informed consent form.

Exclusion Criteria:

* Pregnant women; drug allergy; the patients with serious gastrorrhagia, other peptic ulcers, active bleeding, hepatic insufficiency, heart disease or renal insufficiency; those patients can't tolerate the medicine orally, or participate in other clinical study, or refuse to sign a Informed consent Form.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Hemoglobin | two weeks
  The increased levels of hemoglobin after receiving three different treatment regimens are evaluated in the second week

SECONDARY OUTCOMES:
Reticulocyte | two weeks
  The increased levels of reticulocyte after receiving three different treatment regimens are evaluated in the second week
Hemoglobin | four weeks
  The increased levels of hemoglobin after receiving three different treatment regimens are evaluated in the fourth week
Ferritin | eight weeks
  The increased levels of ferritin after receiving three different treatment regimens are evaluated in the eighth week
adverse events | every two weeks
  The incidence of adverse events every two weeks are assessed, the adverse events include bellyache, diarrhea, constipation, vomiting, nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Qin X Wang, doctorate, Principal Investigator — Huashan Hospital
Locations (1):
- Hushan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brugnara C. A hematologic "gold standard" for iron-deficient states? Clin Chem. 2002 Jul;48(7):981-2. No abstract available. PMID 12089163
- [Background] McCarley P. The KDOQI clinical practice guidelines and clinical practice recommendations for treating anemia in patients with chronic kidney disease: implications for nurses. Nephrol Nurs J. 2006 Jul-Aug;33(4):423-6, 445; quiz 427-8. PMID 17002000
- [Background] Okam MM, Koch TA, Tran MH. Iron deficiency anemia treatment response to oral iron therapy: a pooled analysis of five randomized controlled trials. Haematologica. 2016 Jan;101(1):e6-7. doi: 10.3324/haematol.2015.129114. Epub 2015 Oct 30. No abstract available. PMID 26518747
- [Background] Joseph B, Ramesh N. Weekly dose of Iron-Folate Supplementation with Vitamin-C in the workplace can prevent anaemia in women employees. Pak J Med Sci. 2013 Jan;29(1):47-52. doi: 10.12669/pjms.291.3016. PMID 24353506
- [Background] Parveen N, Ahmad S, Shadab GG. Iron induced genotoxicity: attenuation by vitamin C and its optimization. Interdiscip Toxicol. 2014 Sep;7(3):154-8. doi: 10.2478/intox-2014-0021. Epub 2014 Dec 30. PMID 26109893
- [Background] Rocha Dda S, Capanema FD, Netto MP, de Almeida CA, Franceschini Sdo C, Lamounier JA. Effectiveness of fortification of drinking water with iron and vitamin C in the reduction of anemia and improvement of nutritional status in children attending day-care centers in Belo Horizonte, Brazil. Food Nutr Bull. 2011 Dec;32(4):340-6. doi: 10.1177/156482651103200405. PMID 22590967
- [Derived] Li N, Zhao G, Wu W, Zhang M, Liu W, Chen Q, Wang X. The Efficacy and Safety of Vitamin C for Iron Supplementation in Adult Patients With Iron Deficiency Anemia: A Randomized Clinical Trial. JAMA Netw Open. 2020 Nov 2;3(11):e2023644. doi: 10.1001/jamanetworkopen.2020.23644. PMID 33136134